CLINICAL TRIAL: NCT03693599
Title: Carbetocin Versus Syntometrine for Prevention of Postpartum Hemorrhage in Obese Women Undergoing Elective Cesarean Delivery
Brief Title: Carbetocin Versus Syntometrine in Obese Women Undergoing Elective Cesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: carbetocin
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; syntometrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbetocin (Experimental): 600 women received single 100 µg IV dose of carbetocin diluted in 10 ml of Ringer's lactate solution (Pabal, Ferring Pharmaceuticals Ltd, West Drayton, UK).
  Interventions: Drug: carbetocin
- Syntometrine (Active Comparator): 600 women received one ampoule of syntometrine (Novartis, Basel, Switzerland), which consisted of 5 IU of oxytocin and 500 micrograms of ergometrine diluted in 10 ml of Ringer's lactate solution and was administered intravenously over 2 minutes
  Interventions: Drug: Syntometrine

INTERVENTIONS:
Drug: carbetocin — single 100 µg IV dose of carbetocin diluted in 10 ml of Ringer's lactate solution (Pabal, Ferring Pharmaceuticals Ltd, West Drayton, UK).
  Arms: carbetocin
Drug: Syntometrine — one ampoule of syntometrine (Novartis, Basel, Switzerland), which consisted of 5 IU of oxytocin and 500 microgram of ergometrine diluted in 10 ml of Ringer's lactate solution and was administered intravenously over 2 minutes
  Arms: Syntometrine

SUMMARY:
to compare effectiveness and tolerability of carbetocin versus syntometrine in prevention of Postpartum hemorrhage after cesarean section

DETAILED DESCRIPTION:
A double-blind randomized study conducted on 1200 obese pregnant subjected randomly either to single 100 μg IV dose of carbetocin (600 women) or combination of 5 IU oxytocin and 0.5 mg ergometrine (600 women) after fetal extraction and before placental removal.

Prevention of postpartum haemorrhage (PPH) after cesarean section (CS) had been evaluated by measurement of drop of Hemoglobin and hematocrit, incidence of PPH and number of subjects needed additional oxytocic

ELIGIBILITY:
Inclusion Criteria:

* All participants are at 37 - 40 weeks of gestational age
* Noncomplicated pregnancy.
* obese women with BMI > 30.

Exclusion Criteria:

* Participants with placenta previa,
* coagulopathy,
* preeclamptic
* known sensitivity to carbetocin,oxytocin or methergine were excluded

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of postpartum hemorrhage after CS | 24 hours
  Number of participants experienced massive postpartum hemorrhage

SECONDARY OUTCOMES:
side effects of drugs used | 24 hours
  GIT side effects as nausea , vomiting

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine Cairo university, Giza, Egypt